CLINICAL TRIAL: NCT05111210
Title: Exploration of the Cellular and Molecular Mechanisms in Patients Receiving Biotherapies Targeting the IL-23/IL-17 Axis in Cutaneous Psoriasis
Acronym: Pso23
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-076
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Psoriasis
Keywords: psoriasis; anti-IL-23 therapy; immune responses
MeSH Terms: conditions — Psoriasis | interventions — Blood Specimen Collection; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Gp 1: 10 patients with cutaneous psoriasis: Visits for research are done as part of the care, no visits are added. There is only 1 visit for patients of this group, they will be sampled once with 51 mL of blood before initiation of a biotherapy and some data will be collected
  Interventions: Other: Blood sample; Other: Data collection
- Gp 2: 80 patients with a medical decision to treat cutaneous psoriasis with an anti-IL-23 biologic: Visits for research are done as part of the care, no visits are added. Two visits are planned for this group of patients : before and after initiation of therapy. These patients will be sampled twice with 51 mL of blood. Skin biopsies will be obtained from a subset of 30 patients to analyse the skin transcriptome, before and after treatment with anti-IL-23 biologics Data will be collected at the two timepoints.
  Interventions: Other: Blood sample; Other: Data collection; Other: skin biopsies

INTERVENTIONS:
Other: Blood sample — Blood will be collected in tubes heparinés BD (Vacutainer), homogenised, and immediately transported at room temperature to Institut Pasteur to be further processed
Other: Data collection — collection of socio-demographic, clinical and biological data.
Other: skin biopsies — skin biopsies of 4 mm in diameter. These samples will not be taken on the face or in an area of skin folds
  Groups: Gp 2: 80 patients with a medical decision to treat cutaneous psoriasis with an anti-IL-23 biologic

SUMMARY:
This is a research study involving humans, of the interventional type with minimal risks and constraints (RIPH2). It is a monocentric, non randomized prospective study aiming to better understand the mechanisms of the response to anti-IL-23 biologics in psoriasis patients attending the dermatology department of hospital Cochin (APHP).

DETAILED DESCRIPTION:
The aim of this project is to study the cellular and molecular mechanisms in patients receiving anti-IL-23 biologics as treatment for cutaneous psoriasis, in order to improve the understanding of the role of IL-23/IL-17 axis in this pathology.

This objective is detailed in three specific aims:

* Define the effects of IL-23 on gene expression and cytokine production in innate and adaptive T lymphocytes in patients with skin psoriasis and correlate it with the patient's genotype
* Identify at the single cell level the cells expressing IL-23R and/or producing IL-17 in the skin of patients with skin psoriasis;
* Characterize the in vivo effects of anti-IL-23 therapy on the immune responses of patients with skin psoriasis, by analysing gene expression and protein secretion in whole blood cultures before and after treatment; The secondary objective of this study is to identify mechanisms of non-response to anti-IL-23 therapy in cutaneous psoriasis patients.

The study population to be included are patients affected by cutaneous psoriasis, requiring systemic biological treatment and attended to in the Dermatology Department of the Cochin Hospital. Patients will be divided into two groups: Group 1 patients will participate once before initiation of therapy, Group 2 will participate before and after initiation of anti-IL-23 biologic treatment.

Group 1: 10 patients with cutaneous psoriasis for the phenotypic and transcriptional analyses of T cell populations in peripheral blood. These patients will be sampled once before initiation of biotherapy.

- Group 2: 80 patients with a medical decision to treat cutaneous psoriasis with an anti-IL-23 biologic. These patients will be sampled twice (before and after initiation of therapy), for the analysis of blood immune cell populations using spectral flow cytometry, and immune responses using whole blood cultures. Skin biopsies will be obtained from a subset of 30 patients to analyse the skin transcriptome, before and after treatment with anti-IL-23 biologics.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Adults (>18 years)
* Presenting with cutaneous psoriasis
* Patients have signed an informed consent
* Beneficiary of the health insurance, except for the AME Only for patients of Group 1
* Patients require systemic treatment for psoriasis
* Patients are naïve to biological therapies

Only for patients of Group 2:

* Patients requiring treatment with anti-IL-23 biologics (guselkumab, risankizumab, tildrakizumab) upon referent physician's decision.
* Patients are naïve to biological therapies or have received only one biologic, with a "wash-out" period of at least 4 months

Non inclusion Criteria:

For all :

* Patient is minor
* Patient is pregnant or breastfeeding
* Patient is immunocompromised
* Patient is under legal protection, curatorship, guardianship
* Patient refuses consent
* Patient is unable to comply with study requirements for geographic, social or psychiatric reason.
* Beneficiary of the AME Only for patients of Group 1
* Patient has received biologics Only for patients of Group 2
* Patient has a contraindication to the chosen biotherapy
* Patient has received biologics within the last 4 months
* Patient has been treated with 2 or more biologics
* Patient has already received an anti-IL-23 biologic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population to be included are patients affected by cutaneous psoriasis, requiring systemic biological treatment and attended to in the Dermatology Department of the Cochin Hospital. Patients will be divided into two groups: Group 1 patients will participate once before initiation of therapy, Group 2 will participate before and after initiation of anti-IL-23 biologic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Profiling of open chromatin regions | 7 years
  Profiling of open chromatin regions (ATAC seq), of the transcriptome (RNA-seq), of the genome (genotyping), and of cytokine expression (Luminex technology) in T lymphocytes from patients with cutaneous psoriasis, untreated or treated with IL-23 in vitro
Single cell transcriptome analysis | 7 years
  Single cell transcriptome analysis of skin biopsies from patients with cutaneous psoriasis, before and after anti-IL-23 therapy.
Analysis of the frequencies of MAIT, iNKT, γδ TCR+, CD4+ et CD8+ T cells | 7 years
  Analysis of the frequencies of MAIT, iNKT, γδ TCR+, CD4+ et CD8+ T cells in the peripheral blood of patients with cutaneous psoriasis, before and after initiation of anti-IL-23 treatment to analyse the effect of anti-IL-23 therapy on the immune responses.

SECONDARY OUTCOMES:
Definition of an immune response signature | 7 years
  immune response signature :gene expression, protein secretion or immune cell frequencies that correlates with therapeutic response to anti-IL-23 therapy in cutaneous psoriasis patients.
Identification of epigenetic modifications in cell populations in the skin and/or in circulating immune cells by anti-IL-23 therapy | 7 years
  analyzis of the effects of IL-23 inhibitors on gene expression in specific cell populations isolated from peripheral blood. Particular focis on CD4+ and CD8+ T cells, as well as monocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Lars ROGGE, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided